CLINICAL TRIAL: NCT02960620
Title: A Humanitarian Device Exemption (HDE) Treatment Protocol of TheraSphere® For Treatment of Unresectable Primary or Secondary Liver Neoplasia - HDE #980006
Brief Title: Therasphere for Unresectable Primary or Secondary Liver Neoplasia
Status: No longer available | Type: Expanded Access
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Biocompatibles UK Ltd (Industry); BTG International Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: MCC-15789
Record Dates: First submitted 2016-11-08; First posted 2016-11-09 (Estimated); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Liver Cancer; Liver Neoplasms; HepatoCellular Carcinoma
Keywords: Humanitarian Device Exemption; Liver Disease; HDE #980006
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular; Liver Diseases

INTERVENTIONS:
Device: TheraSphere Treatment — TheraSphere® is delivered into the liver tumor through a catheter placed into the hepatic artery. The hepatic artery provides the main blood supply to the tumor in the liver, whereas the portal vein supplies blood to normal liver parenchyma. TheraSphere® is embolized within the tumor and exerts a local beta radiation radiotherapeutic effect with relatively limited concurrent injury to surrounding normal tissue.

SUMMARY:
This is not a research study. The purpose is to provide supervised access to TheraSphere® therapy at this institution.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be recruited from the patient population referred to the principal clinician for regional liver cancer therapy.
* Potential candidates are those diagnosed with primary or secondary liver neoplasia. The histopathology confirmation criterion may be waived in patients with a radiographically identifiable liver mass, known laboratory or clinical risk factors for cancer or elevated tumor markers and clinical findings. Guidelines from the American Association for the Study of Liver Diseases (AASLD) and the European Association for the Study of the Liver (EASL) describe in detail the approach and algorithm for diagnosing Hepatocellular Carcinoma (HCC).
* Eastern Cooperative Oncology Group (ECOG) Performance Status Score 0 - 2
* Life expectancy ≥ 3 months
* > 4 weeks since prior radiation, surgery or chemotherapy
* Able to comprehend and provide consent in accordance with institutional and federal guidelines

Exclusion Criteria:

* Any other liver therapy planned for cancer treatment
* Uncorrectable flow to the gastrointestinal tract
* Estimated radiation doses to the lungs greater than 30 Gy in a single administration or 50 Gy in multiple administrations
* Significant extrahepatic disease representing imminent life-threatening outcome
* Pregnancy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Junsung Choi, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trials website — https://moffitt.org/clinical-trials-research/